CLINICAL TRIAL: NCT05833698
Title: Acute Uncomplicated Diverticulitis and Conservative Treatment: Accuracy of Inflammatory Indexes for Failure Prediction: Observational Prospective Cohort Study.
Brief Title: Acute Uncomplicated Diverticulitis and Conservative Treatment: Accuracy of Inflammatory Indexes for Failure Prediction: Observational Prospective Cohort Study. (AUDRIP Trial)
Acronym: AUDRIP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Alba Correa Bonito, MD, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: 5072
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Acute Uncomplicated Diverticulitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with failure of conservative treatment
  Interventions: Diagnostic Test: Elevation of NLR
- Patients without failure of conservative treatment
  Interventions: Diagnostic Test: Elevation of NLR

INTERVENTIONS:
Diagnostic Test: Elevation of NLR — Blood test
  Other Names: Elevation of PLR

SUMMARY:
This is an observational multicenter study that will analyse the accuracy of inflammatory indexes as neutrophil-lymphocyte ratio and platelet-lymphocyte ratio, to predict the failure of conservative treatment of patients diagnosed of acute uncomplicated diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18, diagnosed of acute uncomplicated diverticulitis.
* Diagnosis made by CT or ultrasound

Exclusion Criteria:

* Patients younger than 18.
* Patients diagnosed of acute complicated diverticulitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years, diagnosed of acute uncomplicated diverticulitis
Sampling Method: Non-Probability Sample
Enrollment: 2160 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure of conservative treatment with antibiotics | 15th june 2023-31st december 2024
Failure of conservative treatment without antibiotics | 15th june 2023-31st december 2024

SECONDARY OUTCOMES:
Evaluate the accuracy of PLR and NLR as predictors of failure | 15th june 2023-31st december 2024
Analysis of trends in managemente of acute uncomplicated diverticulitis | 15th june 2023-31st december 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided